CLINICAL TRIAL: NCT01772173
Title: Retinal Vessel Measurements as Clinically Useful Predictors in Veterans
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C1084-P
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Diabetes
Keywords: diabetes; computer; retina; vessel; analysis
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Retinal images - vessel parameters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- subjects with diabetes developing hypertension: subjects with diabetes not developing hypertension
  Interventions: Other: Vessel measurements

INTERVENTIONS:
Other: Vessel measurements — Measurement of retinal vessels

SUMMARY:
Diabetic complications are an important source of blindness and mortality among Veterans. Their occurrence is unpredictable because of the highly variable effect of factors such as weight, diet and exercise. Improved prediction of diabetes complications has the potential to improve the care for Veterans with diabetes, especially if this can be done without any extra effort for the Veterans or their caretakers. All Veterans with diabetes in VHA are required to undergo annual retinal photography to screen for current diabetic retinopathy. The investigators have recently developed an automated, precise, fast, novel tool for measuring retinal vessels in these images. Manual measurement of retinal vessels has shown that these can predict future -not current- development of hypertension and also diabetic retinopathy. If the investigators can confirm that their tool can flag those Veterans at increased risk for developing these diabetes complications, this will allow earlier intervention and prevention. Because the tool only uses the images that are being taken anyway, there is no extra effort for either the Veteran or VA staff.

DETAILED DESCRIPTION:
Background: the investigators hypothesize that retinal vessel derived biomarkers, obtained using their automated, precise, fast, novel tool for measuring retinal vessels in retinal images can identify Veterans at increased risk for diabetic retinopathy and hypertension, before any overt signs of retinopathy or increased blood pressure have become apparent. Population studies have shown that changes in arterial and venous diameter are associated with future development of these complications.

Purpose: Determine the potential utility of retinal vessel derived biomarkers, from color fundus photographs, as a non-invasive independent risk factor for diabetic retinopathy (DR) and hypertension in Veterans with diabetes.

Methods: Aim 1. The investigators will evaluate automatically derived retinal vessel parameters (arterial and retinal vessel width and branch relationships) as an early biomarker for future development of hypertension no less than 2 years later, with normal current normal blood pressure. The investigators will compare this biomarker in retinal images from 500 Veterans with diabetes, all of whom did not have hypertension at the time of imaging, for those who were and were not diagnosed with hypertension no more than 3 years later. Aim 2. To evaluate automatically derived retinal vessel parameters as an early biomarker for the risk for development of diabetic retinopathy (defined as transition from less than moderate retinopathy AND no apparent macular edema according to the International Clinical Diabetic Retinopathy and Diabetic Macular Edema Severity Scale) in at risk Veterans with diabetes. The investigators will compare this biomarker in retinal images from a population of 4000 Veterans with diabetes, currently without DR, ~10% of who developed retinopathy no less than two years later while the remainder did not.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with diabetes
* from the Greater LA and Iowa City screening programs
* who were imaged at least 3 years ago for DR screening, and did not have hypertension (AHA definition) at that time

Exclusion Criteria:

* random sample of 500 Veterans with diabetes
* from the Greater LA and Iowa City screening programs
* who were imaged at least 3 years ago for DR screening, and did not have hypertension (AHA definition) at that time

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will identify a random sample of 4500 Veterans with diabetes from the Greater LA and Iowa City screening programs, who were imaged at least 3 years ago for DR screening, and did not have hypertension (AHA definition) at that time
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Area under the Curve of algorithm | 2/1/2016
  AUC of automatically derived retinal vessel parameters (arterial and retinal vessel width and branch relationships) as an early biomarker for future development of hypertension no less than 2 years later, with normal current normal blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Abramoff, MD, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No